CLINICAL TRIAL: NCT03633045
Title: Analysis of Ibrutinib Efficacy and Safety in the Treatment of Chronic Lymphocytic Leukemia Patients in Routine Clinical Practice
Brief Title: Observational Study of Ibrutinib Use in CLL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health (Other)
Responsible Party: Principal Investigator, Conrady Alexandra, Deputy General Director, Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health
Other Study IDs: IB-RU-SCOPE
Record Dates: First submitted 2018-07-20; First posted 2018-08-16 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: CLL, chronic lymphocytic leukemia, ibrutinib
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood. Biobanking of whole blood specimens, collected for routine tests (if available, under separate biobanking informed consent)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
IB-RU-SCOPE is a "routine-clinical practice" oriented cohort observational study of ibrutinib efficacy and safety in approx. 70 patients with chronic lymphocytic leukemia in the Russian Federation

DETAILED DESCRIPTION:
Ibrutinib is approved in Russia for treatment of CLL patients both in first line and in relapsed/refractory setting. There is a discrepancy in reported ibrutinib toxicity profile, efficacy and tolerability between registrational clinical trials and observational studies, which to some extent may be explained by patient selection in the former. IB-RU-SCOPE is a first "routine-clinical practice" oriented cohort observational study of ibrutinib in CLL in Russia. The study is designed to include all previously untreated and relapsed/refractory CLL patients older than 18 years with active disease, who have recently started or are about to start ibrutinib (both as monotherapy and in combination), and to follow them to a minimum of 18 and a maximum of 36 months. The study is being conducted in approx. 10 Russian hematological centers and aims to include approx. 70 CLL patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age older than 18 years.
2. Diagnosis of chronic lymphocytic leukemia, established according to iwCLL criteria (Hallek et al., 2018).
3. Presence of indications for initiating treatment as listed in iwCLL guidelines (Hallek et al., 2018) before start of ibrutinib therapy.
4. Treatment with ibrutinib per instructions for medical use of the drug, approved in the Russian Federation, is planned or this therapy has been started within 7 days before enrolment in the study (date of signing of informed consent). Simultaneously, the patient has not received ibrutinib as one of the previous lines of treatment.
5. Informed consent signed by the patient.

Exclusion Criteria:

1. Presence of contraindications for the use of ibrutinib in accordance with the instructions, approved in the Russian Federation for the medical use of the drug, namely:

* known hypersensitivity to ibrutinib (e.g. with anaphylactic and anaphylactoid reactions);
* pregnancy and the period of breastfeeding;
* age under 18 years;
* severe renal dysfunction (creatinine clearance <30 mL/min), incl. need for hemodialysis;
* severe liver dysfunction (Child-Pugh class C);
* concomitant use with strong inducers of the isoenzyme CYP3A (e.g., carbamazepine, rifampicin, phenytoin and drugs, containing Hypericum perforatum extract);
* concomitant use with warfarin, other vitamin K antagonists, fish oil and vitamin E preparations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males and females with confirmed diagnosis of CLL treated with Ibrutinib
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Frequency of adverse events (including serious adverse events) | 3 years
  In order to evaluate ibrutinib toxicity, all adverse events (AEs), which will occur in study patients, will be collected and analyzed. CTCAE v4.03 criteria and iwCLL criteria will be used for grading of non-hematologic and hematologic AEs, respectively. Frequencies of AEs of all grades will be calculated and reported.
Average duration of treatment with ibrutinib | 3 years
  Time from the first dose of ibrutinib to treatment discontinuation (e.g. due to AEs or CLL progression) will be measured in all study patients. Mean value will be then calculated and reported. This will provide a context, necessary for interpetation of other results (such as toxicity and efficacy measures).
  results (such as toxicity and efficacy measures).
Proportion of patients requiring dose reduction and/or discontinuation of therapy due to causes not related to CLL progression. | 3 years
  In order to evaluate tolerability of ibrutinib in CLL patients in routine clinical practice, all cases of ibrutinib dose reduction and/or drug discontinuation due to causes not related to CLL progression will be collected and analyzed. Proportion of patients, not tolerating full dose of ibrutinib will be then calculated and reported.
Dynamics of QoL indicators assessed by EORTC QLQ-C30 (version 3.0) questionnaire during treatment | 3 yers
  Patients will complete EORTC QLQ-C30 (version 3.0) questionnaires every 3 months during the sudy. Data from questionnaires will be subsequently extracted as numerical values and analyzed according to recommended protocol to estimate changes in patient's quality of life (QoL) during treatment. As a result, either improvement, decline or no change in QoL will be shown

CONTACTS AND LOCATIONS:
Locations (1):
- Almazov FMRC, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No